CLINICAL TRIAL: NCT00789165
Title: A Prospective Trial Of Empiric Quinidine Therapy For Asymptomatic Brugada Syndrome.
Brief Title: Empiric Quinidine for Asymptomatic Brugada Syndrome
Status: Withdrawn | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: International Registry of Asymptomatic Brugada Syndrome (Other)
Responsible Party: Principal Investigator, Dr. Sami Viskin, International RABS director, International Registry of Asymptomatic Brugada Syndrome
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 1297368; No grants at this point
Record Dates: First submitted 2008-11-08; First posted 2008-11-11 (Estimated); Last update posted 2020-02-13 (Actual); Status verified 2020-02

CONDITIONS: Arrhythmia
Keywords: Brugada syndrome; quinidine; Asymptomatic Brugada Syndrome
MeSH Terms: conditions — Arrhythmias, Cardiac; Brugada Syndrome | interventions — Quinidine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Quinidine (Experimental): Patients with type I Brugada electrocardiogram (either spontaneous or following a drug challenge with sodium channel blocker) who never experienced arrhythmia-related symptoms. Patients will receive quinidine therapy at the discretion of the attending physician.
  Interventions: Drug: quinidine
- no therapy (Active Comparator): Patients with asymptomatic Brugada syndrome who opted to receive no therapy following the recommendation of their attending physician
  Interventions: Drug: quinidine; Drug: no therapy

INTERVENTIONS:
Drug: quinidine — quinidine at highest tolerated dose. Expected doses are hydroquinidine 600 - 900 mg daily.
  Other Names: Serecor; Quiniduran
Drug: no therapy — No therapy; this is not a placebo-controlled trial
  Arms: no therapy

SUMMARY:
The purpose of this study is to determine if quinidine therapy (not guided by the results of electrophysiologic studies) will reduce the long-term risk of arrhythmic events in asymptomatic Brugada Syndrome.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with Asymptomatic Brugada syndrome.

   * "Brugada syndrome" is defined as the presence of a Type-I Brugada electrocardiogram [coved ST-segment elevation ≥2 mm (0.2 mV) in V1, V2 or V3] either spontaneously (at rest, in the baseline state or during a febrile episode) or following a standard drug-challenge test (with flecainide, ajmaline, procainamide, or pilsicainide) and recorded either with standard electrode position or with the precordial electrodes placed on the second or third intercostal space. Negative T waves in the precordial leads are not required to define a Type I electrocardiogram.
   * "Asymptomatic patients" will be defined as patients without a history of cardiac arrest, a history of "arrhythmic syncope" or a history of "suspected arrhythmic syncope." Arrhythmic syncope" is a syncope occurring during documented ventricular tachyarrhythmias. "Suspected arrhythmic syncope" is syncope without documented arrhythmias believed to be caused by a tachyarrhythmia based on clinical judgment. In other words, patients with typical vagal syncope will be counted as "asymptomatic" and will be accepted to the registry whereas patients with a clinical history suggesting "syncope other than vagal syncope" will not be accepted to this Registry.
   * Genetic confirmation (identification of a disease-causing mutation) will not be required for establishing the diagnosis of Brugada syndrome but will be recorded when present.
2. Patients with Questionable Brugada Syndrome who are asymptomatic.

   * Patients with "Questionable Brugada Syndrome" are defined as patients with type II or III electrocardiogram who have an inconclusive result during a drug challenge with a sodium channel blocker. "Asymptomatic" is defined as above.
   * Genetic testing will not be required. However, patients with "Questionable Brugada" based on electrocardiographic criteria will be defined as "Patients with Brugada Syndrome" if a disease-causing mutation is identified.

Exclusion Criteria:

1. A history of cardiac arrest, "arrhythmic syncope" or "suspected arrhythmic syncope" (as defined above).
2. Evidence of organic heart disease. The evaluation considered mandatory for excluding heart disease will consist of electrocardiogram, echocardiogram and exercise stress testing. Additional tests will be performed only if clinically indicated.
3. Evidence of non-cardiac disease likely to affect 5-year survival.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2009-12; Primary Completion 2020-02 (Actual); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
Combined endpoint of all cause mortality and spontaneous life-threatening arrhythmias. | Long term (>5 years)

CONTACTS AND LOCATIONS:
Overall Officials: Sami Viskin, M.D., Principal Investigator — Tel Aviv Medical Center
Locations (6):
- Lankenau Institute for Medical Research, Wynnewood, Pennsylvania, United States
- University Medical Centre Mannheim, Mannheim, Germany
- Tel Aviv Medical Center, Tel Aviv, Israel
- University of Pavia and IRCCS Fondazione Policlinico San Matteo, Pavia, Italy
- National Cardiovascular Center, Osaka, Japan
- Academic Medical Centre, Amsterdam, Netherlands